CLINICAL TRIAL: NCT00663806
Title: EXPRESS: Evaluating Cipro XR Patient Response, Education, Safety, and Satisfaction
Brief Title: A Phase IV Study of Cipro XR in Uncomplicated UTI
Acronym: EXPRESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 100534
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Urinary Tract Infections
Keywords: UTI
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Behavioral: Cipro XR (Ciprofloxacin, BAYQ3939)
- Arm 2 (Experimental)
  Interventions: Behavioral: Cipro XR (Ciprofloxacin, BAYQ3939)

INTERVENTIONS:
Behavioral: Cipro XR (Ciprofloxacin, BAYQ3939) — Received Cipro XR (Ciprofloxacin, BAYQ3939) 500 mg once daily for 3 days and brochure about UTI
  Arms: Arm 1
Behavioral: Cipro XR (Ciprofloxacin, BAYQ3939) — Received Cipro XR (Ciprofloxacin, BAYQ3939) 500 mg once daily for 3 days; not given brochure about UTI
  Arms: Arm 2

SUMMARY:
Safety and efficacy of Cipro XR in a naturalistic setting and the effectiveness of an educational brochure. - Women with urinary tract infections were treated with Cipro XR. They were also given a brochure with information about urinary tract infections and later tested on the information.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory women outpatients 18 to 65 years of age with a documented clinical diagnosis of uUTI characterized by dysuria with either urgency or frequency. Women of childbearing age were enrolled only if they were highly unlikely to conceive during the study and were practicing a suitable method of birth control or were at least 1 year postmenopausal.
* Positive leukocyte esterase (>/= 1+) and positive nitrite test using a urine dipstick method of analysis.
* Willing to give written consent.

Exclusion Criteria:

* Pregnant or nursing
* Complicated UTI
* Allergy to Cipro XR

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7614 (Actual)
Dates: Start 2003-02; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
To compare the effect on knowledge of uncomplicated urinary tract infection (uUTI) in patients who were given a disease-directed educational brochure to read versus patients who were not given the brochure. | 3-10 days after start of therapy

SECONDARY OUTCOMES:
To examine the difference between physician and patient perceptions of the symptoms of uUTI. | At baseline visit pre-therapy
To collect data on the clinical efficacy and safety of Cipro XR, 500 mg, PO once daily, for 3 days, in the treatment of uUTI in a naturalistic setting. | 1-3 days after end of therapy for efficacy and up to 30 days for safety

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer